CLINICAL TRIAL: NCT06975904
Title: Effect of Modified Constraint-induced Movement Therapy Combined With Virtual Reality on Mobility in Post-stroke Patients: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/72
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Post Stroke; Mobility; Balance
Keywords: Stroke rehabilitation; Hemiplegia therapy; Motor activity; Gait physiology; Neuroplasticity; Movement disorders rehabilitation; Constraint-Induced Movement Therapy; Virtual reality therapy; Lower extremity pathophysiology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- m-CIMT with Task-Specific Functional Training (Active Comparator): Begin with low-intensity exercises and progress to moderate to high intensity; session will be for about 30 minutes Warm-up for 5 minutes;one minute of rest for every five minutes of exercise For week 1-3: Assisted standing and weight shifting, Heel raises, Toe taps, Supported stepping, Unassisted standing and balance tasks will be used For week 4-6: Progressive stepping exercises, Heel-to-toe standing, Unassisted balance and coordination tasks, Advanced stepping patterns and dynamic balance challenges, Functional tasks like step-ups and lateral steps will be used 5 minutes will be given for cool down
  Interventions: Procedure: m-CIMT with Task-Specific Functional Training
- m-CIMT with VR exer-games by Kinect Xbox 360 (Experimental): Virtual reality workout session will be for about 30 minutes Warm-up exercise will be for 5 minutes including relaxed breathing For week 1-3: Soccer and Space Bubble Pop games will be used For week 4-6: 20,000 Leaks and Rally Ball games will be used 5 minutes will be given for cool down.
  Interventions: Procedure: m-CIMT with VR exer-games by Kinect Xbox 360

INTERVENTIONS:
Procedure: m-CIMT with VR exer-games by Kinect Xbox 360 — Virtual reality workout session will be for about 30 minutes Warm-up exercise will be for 5 minutes including relaxed breathing For week 1-3: Soccer and Space Bubble Pop games will be used For week 4-6: 20,000 Leaks and Rally Ball games will be used 5 minutes will be given for cool down.
  Arms: m-CIMT with VR exer-games by Kinect Xbox 360
Procedure: m-CIMT with Task-Specific Functional Training — Begin with low-intensity exercises and progress to moderate to high intensity; session will be for about 30 minutes Warm-up for 5 minutes;one minute of rest for every five minutes of exercise For week 1-3: Assisted standing and weight shifting, Heel raises, Toe taps, Supported stepping, Unassisted standing and balance tasks will be used For week 4-6: Progressive stepping exercises, Heel-to-toe standing,
  Arms: m-CIMT with Task-Specific Functional Training

SUMMARY:
This study investigates the effectiveness of combining m-CIMT and VR to improve mobility in post-stroke patients. A non-blinded randomized controlled trial will be conducted with 32 participants divided equally into experimental and control groups using purposive sampling. The experimental group will receive m-CIMT with VR training, while the control group will receive m-CIMT with Task-Specific Functional Training. Sessions will be 30 minutes per day, 4 days a week, for 6 weeks. Outcomes will be measured using FMA-LE, BBS, DGI, TUG, and SS-QOL. The study will take place over one year at FFH and FUCP, with ethical approval from ERC FUMC.

ELIGIBILITY:
Inclusion Criteria:

* Sample Selection Criteria

Inclusion Criteria

* Sub-acute and chronic stroke patient >3months
* Males and females of 40-60 years.
* Mini-Mental State Examination score ≥24
* FAC Scale = 3
* Limited spasticity (0,1,1⁺) according to modified Ashworth scale
* Adequate balance and walking ability while wearing the constraint to be eligible to participate in CIMT intervention.

Exclusion Criteria

* Patient with Severe Spasticity and pain
* Patient of Epilepsy, Parkinson's disease and stage 4 arthritis
* Patient with Global Aphasia
* Individuals suffering from unstable angina, symptomatic heart failure, or uncontrolled hypertension
* Patients with any traumatic musculoskeletal injury and surgery of lower limb

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Motor Control | 6 weeks
  Fugl-Meyer Assessment for Lower Extremity (FMA-LE) is a standardized, stroke-specific tool designed to evaluate motor control. It demonstrates excellent reliability (ICC ≥ 0.98) and strong construct validity.
Mobility | 6 weeks
  Time Up and Go test: This test will be used to measure mobility in older adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan